CLINICAL TRIAL: NCT01186276
Title: Dietary Maneuvers to Reduce Production of Colon-Derived Uremic Solutes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SU-07292010-6626; NIH R21AT005123-01A1
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dietary Fiber; Starch

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Corn Starch (Placebo Comparator): Corn starch will serve as the control arm.
  Interventions: Dietary Supplement: Corn starch
- Fiber (Experimental): Fiber will serve as the intervention.
  Interventions: Dietary Supplement: Fiber

INTERVENTIONS:
Dietary Supplement: Fiber — Dietary fiber supplements to be consumed daily for 6 weeks.
  Arms: Fiber
Dietary Supplement: Corn starch — Corn starch to be consumed daily for 6 weeks. This will serve as the control/placebo arm.
  Arms: Corn Starch

SUMMARY:
This study will assess whether dietary fiber supplements can reduce the production of chemicals which are produced by colon bacteria and normally excreted from the body by the kidney, but build up in the body in patients on hemodialysis.

DETAILED DESCRIPTION:
The study procedures will consist of:

* taking a dietary supplement containing either fiber or starch (starch serves as a control for fiber) for six weeks. The fiber dose initially employed will be 30 g/day of high amylose corn and the control starch dose employed will be 30 g/day of waxy corn starch. Supplements which come in dry powder form will be mixed in liquid or food for consumption.
* filling out a food record and a quality of life questionnaire
* keeping a diary of any gi symptoms
* collecting samples of blood, spent dialysate, urine(if the patient still makes urine) and stool.

ELIGIBILITY:
Inclusion Criteria:

* stable dialysis patients able to provide consent.

Exclusion Criteria:-- known g.i. disease

* use of antibiotics for the last two month or expected antibiotic use
* recent hospitalization or other event resulting in instability of food intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Plasma level of p-cresol sulfate | 8 weeks

SECONDARY OUTCOMES:
Caloric intake | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W Meyer, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Satellite Dialysis, Redwood City, California
  - SCVMC, San Jose, California

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148